CLINICAL TRIAL: NCT05742607
Title: Official Title: A Phase II Multicenter, Open Label, Non-randomized Study of Neoadjuvant and Adjuvant Treatment With IPH5201 and Durvalumab in Patients With Resectable, Early-stage (II to IIIA) Non-Small Cell Lung Cancer (MATISSE)
Brief Title: IPH5201 and Durvalumab in Patients With Resectable Non-Small Cell Lung Cancer (MATISSE)
Acronym: MATISSE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Innate Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IPH5201-201
Record Dates: First submitted 2023-02-15; First posted 2023-02-24 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — durvalumab; Carboplatin; Pemetrexed; Drug Therapy

STUDY DESIGN:
Masking Description: Experimental: IPH5201 + durvalumab + chemotherapy
  Patients will receive Neoadjuvant therapy with IPH5201 and durvalumab in addition to standard chemotherapy.
  Following surgery, patients will receive adjuvant treatment with IPH5201 and durvalumab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- IPH5201 + durvalumab + standard chemotherapy (Experimental): Patients will receive Neoadjuvant therapy with IPH5201 and durvalumab in addition to standard chemotherapy.
  Following surgery, patients will receive adjuvant treatment with IPH5201 and durvalumab.
  Interventions: Drug: IPH5201 + durvalumab + standard chemotherapy

INTERVENTIONS:
Drug: IPH5201 + durvalumab + standard chemotherapy — Patients will receive Neoadjuvant therapy with IPH5201 and durvalumab in addition to standard chemotherapy.
  Following surgery, patients will receive adjuvant treatment with IPH5201 and durvalumab.
  Other Names: Durvalumab; MEDI4736, IMFINZI; Carboplatin/Paclitaxel Carboplatin/Paclitaxel, as chemotherapy; Pemetrexed/Cisplatin Pemetrexed/Cisplatin as chemotherapy; Pemetrexed/Carboplatin Pemetrexed/Carboplatin as chemotherapy

SUMMARY:
The study is intended to assess the safety and efficacy of neoadjuvant combination of IPH5201 and durvalumab in addition to standard chemotherapy and adjuvant combination of IPH5201 and durvalumab in untreated patients with resectable, early-stage (stage II to IIIA) non-small cell lung cancer (NSCLC).

DETAILED DESCRIPTION:
This is an open-label, single-arm multicenter study. Eligible patients will be enrolled and will receive IPH5201 + Durvalumab + standard of care chemotherapy before surgery followed by IPH5201 + Durvalumab post-surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed and previously untreated patients with histologically or cytologically documented NSCLC resectable (Stage IIA to Stage IIIA) disease (according to Version 8 of IASLC Staging Manual in Thoracic Oncology 2016.
2. WHO Performance Status or Eastern Cooperative Oncology Group of 0 or 1.
3. Adequate organ and marrow function.
4. Must have a life expectancy of at least 12 weeks.
5. Body weight > 35 kg.
6. Females of childbearing potential should use an acceptable method of contraception from the time of screening throughout the total duration of the study.
7. Negative pregnancy test (serum or urine) for women of childbearing potential.
8. Provision of tumor samples (newly acquired [preferred] or archival tumor tissue [≤ 6 months old]) to confirm Programmed Death-Ligand 1 status, Epidermal Growth Factor Receptor, or Anaplastic Lymphoma Kinase status.
9. Provision of tumor samples appropriate for exploratory biomarker analyses.
10. Patients will be suitable for inclusion if the planned surgery to be performed will be lobectomy, sleeve resection, or bilobectomy, as determined by the attending surgeon based on the baseline findings.
11. A pre- or post-bronchodilator FEV1 of 1.0 L and DLCO > 40% postoperative predicted value.

Exclusion Criteria:

1. Participants with sensitising EGFR mutations or ALK translocations.
2. History of allogeneic organ transplantation.
3. Active or prior documented autoimmune or inflammatory disorders.
4. Uncontrolled intercurrent illness, uncontrolled hypertension, unstable angina pectoris, uncontrolled cardiac arrhythmia, active ILD, serious chronic gastrointestinal conditions associated with diarrhoea, or psychiatric illness/social situations that would limit compliance with study requirement.
5. History of any grade of venous or arterial thromboembolic events including cerebrovascular accident, transient ischemic attack, or unstable angina pectoris within 6 months prior to enrollment.
6. History of another primary malignancy.
7. Patients with small-cell lung cancer or mixed small-cell lung cancer.
8. History of active primary immunodeficiency.
9. Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and tuberculosis testing in line with local practice), hepatitis B (known positive HBsAg result) and HCV. Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody and absence of HBsAg) are eligible. Patients positive for HCV antibody are eligible only if PCR is negative for HCV RNA.
10. Patients who have preoperative radiotherapy treatment as part of their care plan.
11. Patients who require or may require pneumonectomy, segmentectomies, or wedge resections, as assessed by their surgeon, to obtain potentially curative resection of primary tumor.
12. QTc interval ≥ 470 ms (NOTE: If prolonged, then 2 additional ECGs should be obtained and the average QTcF interval should be used to determine eligibility).
13. Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.
14. Any medical contraindication to treatment with chemotherapy as listed in the local labelling.
15. Patients with moderate or severe cardiovascular disease.
16. Any concurrent chemotherapy, investigational product, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable.
17. Receipt of live attenuated vaccine within 30 days prior to the first dose of study interventions.
18. Major surgical procedure (as defined by the Investigator) within 30 days prior to the first dose of study drugs.
19. Prior exposure to immune-mediated therapy.
20. Current or prior use of immunosuppressive medication within 14 days before the first dose of study drugs.
21. Participation in another clinical study with an investigational product administered within 30 days prior to enrolment.
22. Previous study drugs (durvalumab, IPH5201) assignment in the present study.
23. Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 180 days after the last dose of study drugs administration.
24. Involvement in the planning and/or conduct of the study (applies to both company staff and/or staff at the study site).
25. Judgment by the Investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements.
26. Exclusion criteria for participation in the optional (DNA) genetics research component.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-06-23 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Pathological Complete Response (pCR) | 16 weeks after the first dose of study intervention.
  Number of patients with pathological Complete Response (pCR)
Adverse events (AEs) and serious adverse events (SAEs) | Until Day 90 after the last dose of study interventions.
  Number of patients with adverse events (AEs) and serious adverse events (SAEs).

SECONDARY OUTCOMES:
Event-Free Survival (EFS) | Up to approximately 2 years.
  Number of patients experiencing an Event-Free Survival (EFS) event.
Disease Free Survival (DFS) | Up to approximately 2 years.
  Number of patients experiencing a Disease Free Survival (DFS) event (event from surgery onwards).
Surgical resection | Approximately 16 weeks after the first dose of study intervention.
  Number of participants having surgical resection.
Major Pathological Response (mPR) | Approximately 16 weeks after the first dose of study intervention.
  Number of patients with a major Pathological Response (mPR).
Objective Response Rate (ORR) | Up to approximately 4 months adjuvant.
  Number of patients with an Objective Response Rate (ORR).
Overall Survival (OS) | Up to approximately 2 years.
  Overall Survival (OS).
PK of IPH5201 in combination with durvalumab +/- chemotherapy | Up to approximately 4 months adjuvant.
  Serum concentration (PK) of IPH5201 in combination with durvalumab +/- chemotherapy, in patients receiving neoadjuvant and adjuvant treatment.
Anti-study drug antibodies (ADA) | Up to approximately 4 months adjuvant.
  Number of patients with anti-study drug antibodies (ADA).

CONTACTS AND LOCATIONS:
Locations (30):
- United States (6):
  - St. Anthony's Hospital - BayCare Health System, St. Petersburg, Florida
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - University of Chicago Medical Center, Chicago, Illinois
  - Northwell Health Cancer Institute / Center for Novel Cancer Therapeutics, Lake Success, New York
  - Millennium Research & Clinical Development, Houston, Texas
  - UW Carbone Cancer Center - Cancer Connect, Madison, Wisconsin
- France (9):
  - Angers University Hospital Center, Angers
  - University Hospital Center Caen, Caen
  - Hospital Calmette, Lille
  - CHU de Limoges, Limoges
  - Leon Berard Center, Lyon
  - Marseille University Hospital Center - North Hospital, Marseille
  - Rennes University Hospital Center - Hospital Pontchaillou, Rennes
  - Charles Nicolle Hospital, Rouen
  - Gustave Roussy, Villejuif
- Greece (4):
  - Henry Dunant Hospital Center, Athens
  - University General Hospital "Attikon", Athens
  - University General Hospital of Ioannina, Ioannina
  - University General Hospital of Patras, Pátrai
- Hungary (5):
  - Koranyi National Institute of Pulmonology, 14th Department of Pulmonology, Budapest
  - Veszprem County Pulmonology Institute, Farkasgyepű
  - Petz Aladar University Teaching Hospital, Department of Pulmonology, Győr
  - Jasz-Nagykun-Szolnok County Hetenyi Geza Hospital-Clinic, Department of Oncology, Szolnok
  - Pulmonology Institute Torokbalint, Törökbálint
- Poland (6):
  - University Teaching Hospital in Bialystok, 2nd Department of Lung Diseases and Tuberculosis, Bialystok
  - John Paul II Specialist Hospital in Krakow, Krąków
  - Mandziuk Slawomir - Specialist Medical Practice, Lublin
  - Eugenia and Janusz Zeyland Wielkopolskie Centre of Pulmonology and Thoracic Surgery, Poznan
  - Specialist Hospital in Prabuty Sp. z o.o. (LLC), Prabuty
  - Military Institute of Medicine - National Research Institute, Warsaw